CLINICAL TRIAL: NCT06023030
Title: A Post-marketing Non-interventional Study for Upadacitinib in Patients With Moderately to Severely Active Crohn's Disease (CD) in Japan
Brief Title: An Observational Study to Assess Change in Disease Activity and Adverse Events in Adolescent and Adult Participants With Moderate to Severe Active Crohn's Disease (CD) in Japan
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P24-080
Record Dates: First submitted 2023-08-29; First posted 2023-09-05 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; Upadacitinib
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Upadacitinib: Participants will receive upadacitinib as prescribed by their physician according to local label.

SUMMARY:
Crohn's disease (CD) is an incurable chronic inflammatory disorder of the gastrointestinal tract. This study will assess how safe and effective upadacitinib is in treating moderately to severely active CD in real world. Adverse events and change in disease activity will be assessed.

Upadacitinib is a drug approved for the treatment of CD. All study participants will receive upadacitinib as prescribed by their study doctor in accordance with approved local label. Approximately 240 participants will be enrolled in Japan.

Participants will receive upadacitinib as prescribed by their physician according to their routine clinical practice and local label. Participants will be followed for up to 64 weeks.

There is expected to be no additional burden for participants in this trial. Study visits may be conducted on-site or virtually as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with moderately to severely active Crohn's disease (CD).
* Has been prescribed upadacitinib for CD as per most current local approved label after its approval for CD in Japan.
* Within 14 days from the commencement of upadacitinib induction treatment for CD at the participating institution.

Exclusion Criteria:

* Currently participating in another interventional clinical research.
* Participants for whom upadacitinib is contraindicated.
* Has been treated with upadacitinib for CD before and continue treatment with upadacitinib for CD at the participation to this study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and Adult participants with Crohn's disease (CD) in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Drug Related Serious Infections | Up to 64 Weeks
  Pecentage of participants with serious infections.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (101):
- Japan (101):
  - Anjou Kousei Hospital /ID# 261872, Anjo-shi, Aichi-ken
  - Handa City Hospital /ID# 270446, Handa, Aichi-ken
  - Aichi Medical University Hospital /ID# 261871, Nagakute, Aichi-ken
  - Masuko Memorial Hospital /ID# 267420, Nagoya, Aichi-ken
  - Japanese Red Cross Aichi Medical Center Nagoya Daiichi Hospital /ID# 276219, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 275588, Nagoya, Aichi-ken
  - Toyohashi Municipal Hospital /ID# 274975, Toyohashi, Aichi-ken
  - Ieda Hospital /ID# 259754, Toyota-shi, Aichi-ken
  - Hachinohe City Hospital /ID# 264183, Hachinohe, Aomori
  - Tsujinaka Hospital Kashiwanoha /ID# 262648, Kashiwa-shi, Chiba
  - Matsuyama Red Cross Hospital /ID# 266717, Matsuyama, Ehime
  - Uwajima City Hospital /ID# 273444, Uwajima, Ehime
  - Fukuoka University Chikushi Hospital /ID# 262686, Chikushino-shi, Fukuoka
  - Kitakyushu Municipal Medical Center /ID# 276257, Kitakyushu, Fukuoka
  - Tobata Kyoritsu Hospital /ID# 273558, Kitakyushu, Fukuoka
  - Steel Memorial Yahata Hospital /ID# 272713, Kitakyushu, Fukuoka
  - Hidaka Colon Proctology Clinic /ID# 268867, Kurume, Fukuoka
  - Hakuai Clinic /ID# 261876, Kurume-shi, Fukuoka
  - Ashiya Central Hospital /ID# 275324, Onga-gun, Fukuoka
  - Southern Tohoku General Hospital /ID# 270447, Kōriyama, Fukushima
  - Sakura Clinic /ID# 268344, Kakamigahara-shi, Gifu
  - NHO Fukuyama Medical Center /ID# 261873, Fukuyama-shi, Hiroshima
  - JA Hiroshima General Hospital /ID# 264432, Hatsukaichi, Hiroshima
  - Kaisei Clinic /ID# 261883, Hiroshima, Hiroshima
  - Ako-City Hospital /ID# 271276, Ako, Hyōgo
  - Hyogo Prefectural Harima-Himeji General Medical Center /ID# 274528, Himeji, Hyōgo
  - Himeji Chuo Hospital /ID# 272714, Himeji, Hyōgo
  - Itami City Hospital /ID# 276258, Itami, Hyōgo
  - Aoyama Clinic /ID# 262658, Kobe, Hyōgo
  - Kobe City Medical Center General Hospital /ID# 270950, Kobe, Hyōgo
  - Hyogo Medical University Hospital /ID# 267383, Nishinomiya, Hyōgo
  - Kita-Harima Medical Center /ID# 276256, Ono, Hyōgo
  - Tsukuba Endoscopy clinic /ID# 261880, Tsukuba, Ibaraki
  - National Hospital Organization Kanazawa Medical Center /ID# 268820, Kanazawa, Ishikawa-ken
  - Takamatsu Red Cross Hospital /ID# 268823, Takamatsu, Kagawa-ken
  - Maeda Hospital /ID# 275554, Takamatsu, Kagawa-ken
  - Tokai University Hospital /ID# 270949, Isehara, Kanagawa
  - Gokeikai Ofuna Chuo Hospital /ID# 262649, Kamakura-shi, Kanagawa
  - Shimizuogimachi Clinic /ID# 276278, Odawara-shi, Kanagawa
  - Kitasato University Hospital /ID# 276524, Sagamihara-shi, Kanagawa
  - Yokohama Municipal Citizen's Hospital /ID# 267375, Yokohama, Kanagawa
  - Inoue Gastroenterology Clinic /ID# 275555, Yokohama, Kanagawa
  - Saiseikai Yokohama Tobu Hospital /ID# 264186, Yokohama, Kanagawa
  - Chikamori Hospital /ID# 267382, Kochi, Kochi
  - Coloproctology Center Takano Hospital /ID# 268868, Kumamoto, Kumamoto
  - Japanese Red Cross Kyoto Daiichi Hosital /ID# 262660, Kyoto, Kyoto
  - National Hospital Organization Kyoto Medical Center /ID# 265461, Kyoto, Kyoto
  - Mie University Hospital /ID# 262656, Tsu, Mie-ken
  - Yokkaichi Hazu Medical Center /ID# 260140, Yokkaichi-shi, Mie-ken
  - Nagano Municipal Hospital /ID# 262627, Nagano, Nagano
  - Honda Internal Medicine and Endoscopy Clinic /ID# 275628, Nagasaki, Nagasaki
  - Ishida Clinic of IBD and Gastroenterology /ID# 261884, Ōita, Oita Prefecture
  - University of the Ryukyus Hospital /ID# 264430, Ginowan-shi, Okinawa
  - Naha City Hospital /ID# 261875, Naha, Okinawa
  - Seshimo Gastroy & Procto Clinic /ID# 271658, Ibaraki-shi, Osaka
  - Moriguchi Keijinkai Hospital /ID# 268821, Moriguchi, Osaka
  - Kinshukai Infusion Clinic /ID# 261332, Osaka, Osaka
  - National Hospital Organization Osaka National Hospital /ID# 264230, Osaka, Osaka
  - Osaka Metropolitan University Hospital /ID# 273559, Osaka, Osaka
  - Tane General Hospital /ID# 268871, Osaka, Osaka
  - Osaka Rosai Hospital /ID# 267379, Sakai, Osaka
  - Fujita Gastroenterology Hospital /ID# 275410, Takatsuki, Osaka
  - Ohmori Toshihide Gastrointestinal Clinic /ID# 276192, Ageo, Saitama
  - Saitama Medical Center /ID# 270948, Kawagoe, Saitama
  - Tokitokai Tokito clinic /ID# 262661, Saitama-shi, Saitama
  - Tokorozawa Proctogic Hospital /ID# 268870, Tokorozawa, Saitama
  - Kato Clinic /ID# 262650, Hamamatsu, Shizuoka
  - Shizuoka Medical Center /ID# 275551, Shimizu, Shizuoka
  - Shizuoka Aoi Clinic /ID# 267376, Shizuoka, Shizuoka
  - Saigusa Clinic Of Coloproctolo /ID# 275627, Sizuoka-shi, Shizuoka
  - Dokkyo Medical University Hospital /ID# 266710, Mibu, Tochigi
  - Saiseikai Utsunomiya Hospital /ID# 261878, Utsunomiya, Tochigi
  - Juntendo University Hospital /ID# 265452, Bunkyo-ku, Tokyo
  - Ginza Central Clinic /ID# 261881, Chuo-ku, Tokyo
  - Koganei Tsurukame Clinic /ID# 271660, Koganei-shi, Tokyo
  - Ohori IBD Clinic /ID# 261882, Setagaya-ku, Tokyo
  - Shinjuku Tsurukame Clinic /ID# 276485, Shibuya City, Tokyo
  - Tokyo Medical University Hospital /ID# 262683, Shinjuku-ku, Tokyo
  - Tokyo Women'S Medical University Hospital /ID# 274527, Shinjuku-ku, Tokyo
  - The Fraternity Memorial Hospital /ID# 274976, Sumida-ku, Tokyo
  - Yokota Memorial Hospital /ID# 266714, Toyama, Toyama
  - Wakayama Medical University Hospital /ID# 262685, Wakayama, Wakayama
  - Sentohill Hospital /ID# 268869, Ube, Yamaguchi
  - Yamanashi Prefectural Central Hospital /ID# 274526, Kofu, Yamanashi
  - Fukuiken Saiseikai Hospital /ID# 274835, Fukui
  - Fukushima Red Cross Hospital /ID# 275322, Fukushima
  - Gifu University Hospital /ID# 266711, Gifu
  - Japanease Red Cross Society Himeji Hospital /ID# 275590, Himeji
  - Kagoshima IBD Gastroenterology Clinic /ID# 265505, Kagoshima
  - Kuniyoshi Hospital /ID# 271878, Kochi
  - Saga-Ken Medical Centre Koseikan /ID# 274957, Saga
  - Saitama City Hospital /ID# 266716, Saitama
  - Sapporo Kosei General Hospital /ID# 267374, Sapporo
  - Kitasato University Kitasato Institute Hospital /ID# 268345, Tokyo
  - Tokyo Yamate Medical Center /ID# 275591, Tokyo
  - Teikyo University Hospital /ID# 274525, Tokyo
  - Teikyo University Hospital /ID# 274977, Tokyo
  - Municipal Toyonaka Hospital /ID# 266712, Toyonaka
  - Japanese Red Cross Society - Wakayama Medical Center /ID# 268822, Wakayama
  - Yamagata Prefectural Central Hospital - Yamagata /ID# 268819, Yamagata
  - Yamaguchi Red Cross Hospital /ID# 267381, Yamaguchi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P24-080